CLINICAL TRIAL: NCT03550131
Title: Aging With Pride: Innovations in Dementia Empowerment and Action
Brief Title: Innovations in Dementia Empowerment and Action
Acronym: IDEA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Karen Fredriksen Goldsen, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00003076; 1R01AG055488-01A1 (NIH)
Record Dates: First submitted 2018-04-06; First posted 2018-06-08 (Actual); Results first posted 2024-07-25 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease; Dementia; Mild Cognitive Impairment; Parkinson Disease Dementia; Lewy Body Dementia; Vascular Dementia
Keywords: LGBT
MeSH Terms: conditions — Alzheimer Disease; Dementia; Cognitive Dysfunction; Lewy Body Disease; Dementia, Vascular | interventions — Amyloid beta-Protein Precursor

STUDY DESIGN:
Intervention Model Description: This study will utilize a 2-group randomized controlled trial design including 2 pre-intervention and 4 post-intervention assessments. The comparator group (standard intervention) will have 112 caregiver-care receiver dyads, and the experimental group (personalized intervention) will have 113 caregiver-care receiver dyads.
Who Masked: Participant
Masking Description: Participants receiving intervention will not be informed whether it is the standard or personalized treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard intervention (Active Comparator): Reducing Disabilities in Alzheimer's Disease (RDAD):
  9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Interventions: Behavioral: Reducing Disabilities in Alzheimer's Disease (RDAD)
- Personalized intervention (Experimental): Innovations in Dementia Empowerment and Action (IDEA):
  9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Interventions: Behavioral: Innovations in Dementia Empowerment and Action (IDEA)

INTERVENTIONS:
Behavioral: Innovations in Dementia Empowerment and Action (IDEA) — The IDEA intervention has the same exposure to treatment as the RDAD intervention. The behavioral component of the treatment manual is adapted to incorporate 3 risk factors that are empirically known to affect midlife and older LGBT populations.These include: 1) identity management; 2) stigma-related adverse/traumatic life events; and 3) lack of social support. All other aspects of the treatment are preserved.
  Other Names: Personalized RDAD
  Arms: Personalized intervention
Behavioral: Reducing Disabilities in Alzheimer's Disease (RDAD) — The RDAD intervention includes behavioral management training for caregiver and activities and exercise training for caregiver and care receiver.
  Other Names: Standard RDAD
  Arms: Standard intervention

SUMMARY:
The lack of efficacious research-based interventions for such vulnerable older adults with Alzheimer's disease and related dementias (AD/RD) and their caregivers (CGs) is a significant public health problem. Caregiving of sexual/gender minority older adults with AD/RD is of concern due to social stigma, marginalization, and isolation, which may be barriers to sustaining caregiving. It is necessary and timely to translate evidence-based culturally adaptable interventions for this underserved and stigmatized population. Reducing Disability in Alzheimer's Disease (RDAD) has been evaluated in a randomized controlled trial and has shown to successfully train community-dwelling CR (care receiver)-CG dyads to increase the physical activity and functioning of individuals with AD/RD and their CGs and to teach CGs techniques for managing behavioral symptoms of CRs. RDAD consequently decreases stress of CGs, delays institutionalization of CRs, and increases health related quality of life (HRQOL) of CRs and CGs. Thus, this study will evaluate the effect of the standard RDAD among lesbian, gay, bisexual, and transgender (LGBT) CRs with AD/RD and their CGs, and this study will test a personalized intervention tailored to better respond to distinct risks experienced by CGs and LGBT CRs with AD/RD, addressing unique sexual/gender minority CG risk factors (e.g., identity management, stigma-related adverse or traumatic life events, and lack of social support).

DETAILED DESCRIPTION:
We will address the following aims:

Aim 1. Test the translation and enhancement of intervention designed to increase physical activities of older adult care receivers (CRs) with AD/RD and their CGs. Aim 2. Evaluate the short- and long-term effect of the standard and personalized intervention on primary (physical activity and functioning; perceived stress for CGs; independence/residential status (institutionalization) for CRs) and secondary outcomes (HRQOL; depressive symptomatology; behavioral disturbances for CRs). Aim 3. Test the moderating roles of CR-CG characteristics, including type of CR-CG relationship, sex, and severity of CR AD/RD, on the treatment effect of the standard and personalized intervention.

ELIGIBILITY:
Inclusion criteria for care receiver

* Age at enrollment is 50 years of age or older
* Have dementia, (e.g., Alzheimer's disease, mild cognitive impairment, Vascular dementia, Parkinson's disease, Lewy Body dementia) or memory loss significant enough to affect daily activities
* Living in the community, not in a care facility.
* Living in the U.S.
* Either the care receiver or care giver must self-identify as LGBT (or sexual or gender non-binary or same sex sexual behavior)

Inclusion criteria for care giver

* Provide care to the care recipient with dementia.
* Willing to spend 30 minutes daily for study activities (or coordinate for someone to.)
* Unpaid
* Live in the community, not in a care facility
* Living in the U.S.

Neither care receiver nor caregiver:

* Has known terminal illness (with death anticipated within the next 12 months)
* Was hospitalized for a psychiatric disorder in the 12 months prior to baseline
* Is currently suicidal or having major hallucinations or delusions
* Plans to move to long term care setting within 6 months of enrollment.
* Has any physical limitations/chronic conditions preventing participation in an exercise program.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2018-12-05 (Actual); Primary Completion 2023-05-16 (Actual); Study Completion 2023-05-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Fredriksen-Goldsen, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

REFERENCES:
- [Derived] Fredriksen-Goldsen KI, Teri L, Kim HJ, Jones-Cobb B, LaFazia D, McKenzie G, Petros R, Jung H, Oswald AG, Hoy-Ellis C, Emlet C. Innovations in Dementia Empowerment and Action: RCT for Underserved Communities. J Am Geriatr Soc. 2026 Jan;74(1):119-131. doi: 10.1111/jgs.70189. Epub 2025 Dec 12. PMID 41387197

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from multiple sources using a multifaceted approach, including direct referrals from community agencies providing aging and health services using presentations, flyers, newsletters, and social media.
Pre-assignment Details: A total of 161 dyad pairs (i.e., a person with dementia and their care partner) were enrolled and randomly assigned to either the personalized or standard arm.
Groups:
- Personalized Intervention: Innovations in Dementia Empowerment and Action (IDEA):
  9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Innovations in Dementia Empowerment and Action (IDEA): The IDEA intervention has the same exposure to treatment as the RDAD intervention. The behavioral component of the treatment manual is adapted to incorporate 3 risk factors that are empirically known to affect midlife and older lesbian, gay, bisexual, and transgender (LGBT) populations.These include: 1) identity management; 2) stigma-related adverse/traumatic life events; and 3) lack of social support. All other aspects of the treatment are preserved.
- Standard Intervention: Reducing Disabilities in Alzheimer's Disease (RDAD):
  9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Reducing Disabilities in Alzheimer's Disease (RDAD): The RDAD intervention includes behavioral management training for caregiver and activities and exercise training for caregiver and care receiver.
Period: Overall Study
Arm/Group | Personalized Intervention | Standard Intervention
Started | 162 (A dyad consists of a care recipient with dementia and their care partner. The personalized arm enrolled 81 dyads, resulting in 162 participants.) | 160 (A dyad consists of a care recipient with dementia and their care partner. The personalized arm enrolled 80 dyads, resulting in 160 participants.)
Baseline, CR | 80 | 76
Baseline, CP | 80 | 76
6 Week (Pre-Treatment), CR | 70 | 71
6 Week (Pre-Treatment), CP | 70 | 71
13 Week (Post-treatment), CR | 57 | 63
13 Week (Post-treatment), CP | 57 | 63
30 Week Follow up, CR | 53 | 61
30 Week Follow up, CP | 53 | 61
13 Month Follow up, CR | 48 | 49
13 Month Follow up, CP | 48 | 49
Completed | 96 | 98
Not Completed | 66 | 62
Not completed — Lost to Follow-up | 16 | 24
Not completed — Withdrawal by Subject | 36 | 28
Not completed — Illness of dyad member | 10 | 2
Not completed — Death of person with dementia | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Personalized Intervention: Innovations in Dementia Empowerment and Action (IDEA):
  9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Innovations in Dementia Empowerment and Action (IDEA): The IDEA intervention has the same exposure to treatment as the RDAD intervention. The behavioral component of the treatment manual is adapted to incorporate 3 risk factors that are empirically known to affect midlife and older LGBT populations.These include: 1) identity management; 2) stigma-related adverse/traumatic life events; and 3) lack of social support. All other aspects of the treatment are preserved.
- Total: Total of all reporting groups
Arm/Group | Personalized Intervention | Standard Intervention | Total
Number analyzed (Participants) | 80 | 76 | 156
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The overall number includes both care recipients and care partners.
  years
    Care recipient (CR) | 69.36 (10.11) | 72.19 (8.26) | 70.75 (9.32)
    Care partner (CP) | 62.15 (13.04) | 62.03 (13.34) | 62.09 (13.15)
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: The overall number includes both care recipients and care partners.
  Participants
    Care recipient (CR): Women | 47 | 45 | 92
    Care recipient (CR): Men | 33 | 28 | 61
    Care recipient (CR): Diverse | 0 | 3 | 3
    Care partner (CP): Women | 45 | 38 | 83
    Care partner (CP): Men | 30 | 32 | 62
    Care partner (CP): Diverse | 5 | 6 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number includes both care recipients and care partners.
  Participants
    Care recipient (CR): Hispanic or Latino | 9 | 4 | 13
    Care recipient (CR): Not Hispanic or Latino | 71 | 72 | 143
    Care recipient (CR): Unknown or Not Reported | 0 | 0 | 0
    Care partner (CP): Hispanic or Latino | 7 | 5 | 12
    Care partner (CP): Not Hispanic or Latino | 73 | 71 | 144
    Care partner (CP): Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The overall number includes both care recipients and care partners.
  Participants
    Care recipient (CR): American Indian or Alaska Native | 0 | 1 | 1
    Care recipient (CR): Asian | 0 | 0 | 0
    Care recipient (CR): Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
    Care recipient (CR): Black or African American | 7 | 3 | 10
    Care recipient (CR): White | 67 | 68 | 135
    Care recipient (CR): More than one race | 4 | 3 | 7
    Care recipient (CR): Unknown or Not Reported | 2 | 0 | 2
    Care partner (CP): American Indian or Alaska Native | 0 | 3 | 3
    Care partner (CP): Asian | 3 | 3 | 6
    Care partner (CP): Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Care partner (CP): Black or African American | 4 | 3 | 7
    Care partner (CP): White | 62 | 58 | 120
    Care partner (CP): More than one race | 10 | 6 | 16
    Care partner (CP): Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity of Care Recipient
Description: Measured by the days of aerobic activity for at least 30 minutes in the past week with higher numbers indicating more days of activity.
Time Frame: Baseline, 6 weeks(pre-treatment), 13 weeks(post-treatment), 30 weeks, 13 months
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Personalized Intervention | Standard Intervention
Number analyzed (Participants) | 80 | 76
days
  Baseline | 3.20 (2.56) | 2.76 (2.53)
  6 weeks | 3.01 (2.66) | 2.66 (2.53)
  13 weeks | 3.81 (2.40) | 3.79 (2.54)
  30 weeks | 3.67 (2.67) | 3.21 (2.60)
  13 months | 2.96 (2.51) | 2.96 (2.51)

2. Secondary Outcome: Depression of Care Partner: Center for Epidemiological Studies-Depression Scale (CESD-10)
Description: Assessed using the summed score on the 10-item Center for Epidemiological Studies-Depression Scale (CESD-10). Range of scores 0-27 with higher scores indicating higher levels of depression.
Time Frame: Baseline, 6 weeks(pre-treatment), 13 weeks(post-treatment), 30 weeks, 13 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Intervention | Standard Intervention
Number analyzed (Participants) | 80 | 76
score on a scale
  Baseline | 7.38 (5.45) | 6.98 (5.57)
  6 weeks | 6.76 (6.29) | 6.95 (5.01)
  13 weeks | 5.63 (5.58) | 6.38 (5.22)
  30 weeks | 6.43 (5.98) | 7.21 (4.62)
  13 months | 5.23 (5.58) | 5.70 (6.22)

3. Secondary Outcome: Quality of Life in Alzheimer's Disease, Care Recipient
Description: Quality of life was evaluated using the summed score of the Quality of Life in Alzheimer's Disease (QOL-AD), a 13-item measure. Range of scores 13-52 with higher scores equal better quality of life.
Time Frame: Baseline, 6 weeks(pre-treatment), 13 weeks(post-treatment), 30 weeks, 13 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Intervention | Standard Intervention
Number analyzed (Participants) | 80 | 76
score on a scale
  Baseline | 33.29 (6.46) | 34.71 (7.13)
  6 weeks | 33.94 (5.98) | 34.07 (7.05)
  13 weeks | 36.49 (6.42) | 35.37 (6.87)
  30 weeks | 35.46 (6.12) | 34.79 (6.80)
  13 months | 33.94 (7.31) | 35.37 (6.82)

4. Secondary Outcome: Memory-Related Disturbance, Care Recipient
Description: Assessed using mean scores on the memory-related subscale (7 items) of the 24-item Revised Memory and Behavior Problem Checklist (RMBPC). Ranges 0 -3. Higher scores indicate higher memory-related behavioral disturbances.
Time Frame: Baseline, 6 weeks(pre-treatment), 13 weeks(post-treatment), 30 weeks, 13 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Intervention | Standard Intervention
Number analyzed (Participants) | 80 | 76
score on a scale
  Baseline | 1.24 (0.78) | 1.19 (0.72)
  6 weeks | 1.21 (0.80) | 1.15 (0.73)
  13 weeks | 1.10 (0.80) | 1.10 (0.76)
  30 weeks | 1.21 (0.85) | 1.14 (0.79)
  13 months | 1.29 (0.93) | 1.14 (0.84)

5. Secondary Outcome: Physical Functioning of Care Recipient: Medical Outcomes Study 36-Item Short Form (SF-36)
Description: Physical functioning was assessed using the mean score of the Physical Functioning subscale of the Medical Outcomes Study 36-Item Short Form (SF-36), consisting of 10 items asking about degree to which health status limits activities including walking, climbing, lifting, and bathing or dressing oneself. The summary score ranges from 0 to 100. Higher scores indicate higher physical functioning.
Time Frame: Baseline, 6 weeks(pre-treatment), 13 weeks(post-treatment), 30 weeks, 13 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Intervention | Standard Intervention
Number analyzed (Participants) | 80 | 76
score on a scale
  baseline | 58.65 (28.37) | 58.46 (31.04)
  6 weeks | 58.15 (28.98) | 59.16 (30.19)
  13 weeks | 59.95 (28.40) | 61.24 (31.70)
  30 weeks | 58.17 (30.13) | 57.79 (32.00)
  13 months | 59.79 (29.98) | 57.45 (30.62)

6. Secondary Outcome: Perceived Stress of Care Partner
Description: Assessed with mean scores of the 4-item Perceived Stress Scale. The summary score ranges from 0 to 4. Higher scores indicate more stress.
Time Frame: Baseline, 6 weeks (Pre-treatment), 13 weeks (Post-treatment), 30 weeks, 13 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Personalized Intervention | Standard Intervention
Number analyzed (Participants) | 80 | 76
score on a scale
  Baseline | 2.39 (0.28) | 2.42 (0.25)
  6 weeks | 2.46 (0.27) | 2.44 (0.22)
  13 weeks | 2.44 (0.29) | 2.46 (0.30)
  30 weeks | 2.43 (0.29) | 2.43 (0.26)
  52 weeks | 2.41 (0.23) | 2.41 (0.25)

ADVERSE EVENTS:
Time Frame: 56 weeks
Groups:
- Personalized Intervention, Care Recipient; Personalized Intervention, Care Partner: Innovations in Dementia Empowerment and Action (IDEA): 9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Innovations in Dementia Empowerment and Action (IDEA): The IDEA intervention has the same exposure to treatment as the RDAD intervention. The behavioral component of the treatment manual is adapted to incorporate 3 risk factors that are empirically known to affect midlife and older LGBT populations. These include: 1) identity management; 2) stigma-related adverse/traumatic life events; and 3) lack of social support. All other aspects of the treatment are preserved.
- Standard Intervention, Care Recipient; Standard Intervention, Care Partner: Reducing Disabilities in Alzheimer's Disease (RDAD): 9 60-minute virtual sessions for 6 weeks and 4 15-minute follow-up phone sessions for 4 months
  Reducing Disabilities in Alzheimer's Disease (RDAD): The RDAD intervention includes behavioral management training for caregiver and activities and exercise training for caregiver and care receiver.
Arm/Group | Personalized Intervention, Care Recipient | Personalized Intervention, Care Partner | Standard Intervention, Care Recipient | Standard Intervention, Care Partner
All-Cause Mortality (participants affected / at risk) | 2/80 | 0/80 | 4/76 | 0/76
Serious Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/76 | 0/76
Other Adverse Events (participants affected / at risk) | 0/80 | 0/80 | 0/76 | 0/76

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2021-08-26): https://cdn.clinicaltrials.gov/large-docs/31/NCT03550131/Prot_SAP_000.pdf
  • Informed Consent Form: Care Partner (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03550131/ICF_001.pdf
  • Informed Consent Form: Care Recipient (2021-07-09): https://cdn.clinicaltrials.gov/large-docs/31/NCT03550131/ICF_002.pdf